CLINICAL TRIAL: NCT06648161
Title: Impact of Using a Mirror in the Second Stage of Labor on Childbirth Duration and Experience
Brief Title: Using a Mirror in the Second Stage of Labor: Effects on Duration and Birth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Resmiye Ozdilek, Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Suzi-02
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Labor Stage, Second
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): In the second stage of labor, the birth mirror will be used to allow the mother to see her own perineum.
  Interventions: Other: Labor Mirror
- Control (No Intervention): During the birth process, she will receive routine midwifery care and no intervention will be made.

INTERVENTIONS:
Other: Labor Mirror — The labor mirror used in the second stage of labor allows the mother and midwife to observe the descent and birth of the baby during vaginal delivery and provides instant visualization of progress for the mother and midwife, especially in water births or water births
  Arms: Experiment

SUMMARY:
This study aims to investigate the impact of using a labor mirror during the second stage of labor on both the duration of labor and the mother's overall experience. The main questions it aims to answer are:

* Does using a labor mirror in the second stage of labor affect the duration of labor?
* Does the use of a labor mirror in the second stage of labor affect women's total birth experience scale score? To assess the effect of using a birth mirror during the second stage of labor on the duration of labor and mothers' satisfaction with labor, the researchers will give one group a birth mirror and the other group will receive normal midwifery care.
* In the second stage of labor, the birth mirror will be positioned so that the woman can see the progress of the baby as she pushes (lithotomy position).
* Within 24 hours after delivery, mothers will complete the Birth Experience Scale and an opinion form about the use of the mirror.
* The control group will not receive any intervention.

DETAILED DESCRIPTION:
Childbirth is one of the most significant experiences in a woman's life. The second stage of labor, when the cervix is fully dilated and the baby moves through the birth canal, is a crucial phase. Various techniques and tools are used during this stage to assist delivery, one of which is the labor mirror. This tool allows the mother to visually observe the perineum and monitor the progress of labor, especially in water births. Both handheld and bed-mounted options are available, usually made of acrylic, and they can have adjustable angles for better visualization.

The use of a labor mirror offers several benefits. It enables real-time monitoring of the birthing process, allowing midwives to make timely interventions. More importantly, it helps mothers feel more involved in the birth, boosting their confidence and motivation, especially when they see the baby's head. This can lead to more controlled pushing and potentially shorten the duration of labor.

In summary, the labor mirror can enhance the birth experience by allowing mothers to participate actively and by providing emotional support, which may reduce the length of the second stage of labor. However, its use is not widespread in Turkey. This study aims to investigate the impact of using a labor mirror during the second stage of labor on both the duration of labor and the mother's overall experience.

ELIGIBILITY:
Inclusion Criteria:

* between 38-42 weeks of gestation,
* had a healthy fetus,
* had no perinatal and obstetric risk,
* did not have prolonged trauma,
* could understand and speak Turkish

Exclusion Criteria:

* preterm labor onset,
* premature rupture of membranes,
* epidural analgesia,
* amniotic fluid with meconium,
* fetal risk
* intervention delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experiment | Control
Started | 61 | 61
Completed | 61 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experiment | Control | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 61 | 122
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.82 (5.35) | 25.92 (5.02) | 26.37 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 61 | 61 | 122
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 61 | 61 | 122
Gestational Week at Admission [Mean (Standard Deviation); unit: Weeks] — Mean gestational week at admission was calculated for each study group prior to intervention. This measure indicates the pregnancy week based on the last menstrual period and/or ultrasound assessment at the time of hospital admission for labor. Units are expressed in completed weeks.
  Weeks | 39.21 (1.20) | 39.33 (1.21) | 39.27 (1.20)

OUTCOME MEASURES:

1. Primary Outcome: Childbirth Experience Questionnaire (CEQ) Total Score
Description: The Childbirth Experience Questionnaire (CEQ) is a validated scale measuring women's birth experiences. It has 22 items across 4 subscales. Total score is the sum of all items converted to a 1-4 scale, yielding a range of 22-88. Higher scores indicate a more positive childbirth experience.
Time Frame: Within 24 hours postpartum
Population: The analysis included women who completed the Childbirth Experience Questionnaire within 24 hours after delivery. Participants who withdrew or had incomplete data were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experiment | Control
Number analyzed (Participants) | 61 | 61
units on a scale | 73.85 (9.76) | 70.22 (9.60)

2. Secondary Outcome: Duration of the Second Stage of Labor
Description: The duration of the second stage of labor was compared between the experimental and control groups to assess the impact of labor mirror use.
Time Frame: During the second stage of labor, within the birth process
Population: All participants who completed the second stage of labor with recorded time data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Experiment | Control
Number analyzed (Participants) | 61 | 61
Minutes | 12.52 (4.53) | 19.48 (5.58)

ADVERSE EVENTS:
Time Frame: From the onset of the second stage of labor until delivery completion and during the first 24 hours postpartum.
Description: No adverse or serious adverse events were observed or reported during the study. Adverse events were monitored during the second stage Participants were monitored for any adverse or serious adverse events during the second stage of labor, delivery, and the first 24 hours postpartum. Standard obstetric observation protocols were followed. No free-text repetition of numerical results is provided; all event counts are presented in the data tables.
Arm/Group | Experiment | Control
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT06648161/Prot_SAP_000.pdf